CLINICAL TRIAL: NCT07367867
Title: Inflammation in HIV/AIDS-InflammAIDS: an Observational Multicenter Cohort Study Protocol
Brief Title: Inflammation in HIV/AIDS-InflammAIDS
Acronym: InflammAIDS
Status: Completed | Type: Observational
Sponsor: Universidad de Magallanes (Other)
Collaborators: University of Chile (Other)
Responsible Party: Principal Investigator, Marcelo A. Navarrete Signorile, Principal Investigator, Universidad de Magallanes
Other Study IDs: ATE220016; ATE220016 (Other Grant/Funding Number: Concurso Anillos de Investigación ANID)
Record Dates: First submitted 2025-08-19; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: HIV; Metabolic Syndrome; Molecular Biology; Flow Cytometry; Sequence Analysis; Single Cell Sequencing Technology; Microbiome
Keywords: interdisciplinary group of researchers; PLWH; metabolic syndrome; Chile; HIV; Biobank standards
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — 1) Plasma samples: Venous samples will be collected in EDTA-containing tubes. They will be centrifuged for 15 minutes at 1000 g and then fractionated into blood cells and plasma. Plasma will be aliquoted and stored for further processing. 2) Isolation of PBMCs: PBMCs will be obtained from whole blood samples. The untouched PBMCs will be collected into a tube and mixed with cryopreservation medium to avoid cell lysis. Cells will be frozen in liquid nitrogen and transported to be stored until used. 3) Stool samples: A stool sample will be collected. Tubes will be then stored until further processing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- InflammAIDS cohort is a PLWH cohort with and without metabolic syndrome: The InflammAIDS cohorts is a PLWH cohort from different centers of Santiago and Punta Arenas, including Fundación Arriarán, Hospital Clínico de Magallanes and Hospital del Salvador. These cohorts include men and women, from adolescence to adulthood and senior patients living with HIV under suppressive ART and presenting or not metabolic syndrome. Importantly, the project also have access to a pediatric cohort, including children living with HIV and without metabolic syndrome. A group of HIV negative individuals with and without metabolic syndrome will also be invited to participate to be used as controls when required.

SUMMARY:
The human immunodeficiency virus/acquired immunodeficiency syndrome (HIV/AIDS) pandemic still represents a major public health problem with 41 million people currently living with HIV worldwide. Indeed, the advent of antiretroviral therapy (ART) has largely decreased morbidity and mortality associated with HIV/AIDS. Nevertheless, ART is not able to eradicate the virus and, therefore, the management of HIV/AIDS involves a long-term treatment. The persistence of an HIV reservoir is associated with a chronic status of immune activation and inflammation, exacerbating damage in tissues. Consequently, the immunological status of people living with HIV (PLWH) is reminiscent to what is observed in immunosenescence, predisposing them to the development of the so-called non-AIDS defining diseases (NADE), which correspond to conditions commonly observed in aging such as metabolic syndrome, cardiovascular diseases, diabetes, neurocognitive disorders, and non-HIV associated cancers, amongst others. The investigators estimate that more than a half of Chilean patients present metabolic syndrome, a well characterized risk factor including cardiovascular disease , type 2 diabetes and death in the general population but especially in PLWH. The Anillo Inflammation in HIV/AIDS (InflammAIDS) brings together an interdisciplinary group of researchers from life and medical sciences working at public universities and hospitals with the aim of investigating the immune, inflammatory and virological signatures of PLWH with and without metabolic syndrome in Chile and how they influence the clinical outcome of the patients. To accomplish our objectives, the researchers group will first establish a prospective cohort of PLWH, with and without metabolic syndrome, across relevant lifetime periods (childhood, adulthood, and elderly) and will generate the first Chilean collection of samples from the participants of this clinical cohort with Biobank standards, generation standardized and high-quality sample and data collection. These cohorts will be analyzed combining state-of-the-art methodologies such as single-cell RNA sequencing, multiparametric flow cytometry, xMap® Luminex, mass spectrometry and Oxford Nanopore Technologies sequencing together with classical biochemical, molecular, and cellular biology, virological and immunological analyses, determining the immune, inflammatory and virological state associated to the clinical condition of our patients.

DETAILED DESCRIPTION:
Human immunodeficiency virus (HIV), as the etiological agent of AIDS (Acquired immunodeficiency syndrome) in humans. Forty years since HIV/AIDS emergence, HIV still represents an important threat to the human population and a major public health problem. According to the last report from UNAIDS, close to 80 million individuals have been infected by HIV and 36 million have died by an AIDS-related disease since the beginning of the pandemic. Chile has not been exempted of the HIV/AIDS syndemic, experiencing an important increase in HIV infections from 2,982 confirmed cases by 2010 to 4,446 and 5,031 new confirmed infections in 2020 and 2021, respectively, despite the restrictions in diagnosis imposed by the COVID-19 pandemic. Although most of the diagnosed individuals are under suppressive treatment, an important 45% of the new HIV infections in Chile are detected at late stages of infection (mostly at the AIDS stage), a condition associated with a lower quality of life. Moreover, while 70% of the PLWH in Chile correspond to adults aged 15-49, there is a non-negligible number of children and adolescents living with HIV, who acquired infection both vertically or horizontally, as well as an increasing population aged 50 and over. Importantly, the estimation that more than a half of the patients visiting the chilean health centers present metabolic syndrome, a known risk factor for other conditions associated with a poor clinical outcome including cardiovascular disease (CVD), type 2 diabetes and death. The advent of combined antiretroviral therapy (ART) has revolutionized prognosis of PLWH by decreasing morbidity and mortality associated with HIV infection. The success of ART in suppressing circulating viral RNA levels (viral load) below the limits of detection is due to the inhibition of active viral replication, which mainly occurs in activated CD4+ T-cells. However, despite an undetectable viral load in plasma, the discontinuation of ART leads to viral rebound within weeks due to the so-called latent reservoir, (memory CD4+ T-cells), which carry integrated, transcriptionally silenced, replication-competent proviral DNA. Moreover, resting memory CD4+ T-cells bypass immune surveillance, are refractory to the effects of ART, are long-lived and undergo clonal expansion, making them an ideal niche for viral persistence. The latent reservoir is established within hours following infection and persists in different anatomical niches (including lungs, gut-associated lymphoid tissue, lymph nodes, central nervous system and adipose tissue), despite successful viral suppression by ART and, upon an activation stimulus, latency is reversed leading to viral rebound with subsequent clinical deterioration. Monocytes and macrophages and their role in HIV replication and persistence CD4+ T-cells are not the only cell type in which HIV is able to establish a latent reservoir and persist for prolonged periods. Indeed, there is increasing evidence showing that monocyte-derived macrophages (MDM), including different tissue-resident macrophages, contain HIV DNA, RNA, and proteins in individuals under suppressive ART and M-tropic HIV can be detected upon ART interruption. Monocytes also play a critical role in HIV dissemination as they migrate to seed multiple tissues during infection. Moreover, macrophages play a critical role during untreated infection, particularly at late stages when CD4+ T cells are depleted, being the principal drivers of viremia. In contrast to MDM, which corresponds to terminally differentiated non-dividing cells, microglia (the CNS resident macrophages) undergo self-renewal and are maintained in the brain for the entire life. Therefore, HIV- infected macrophages and microglia also serve as long-term tissue reservoirs contributing to viral persistence and tissue damage even under suppressive ART. Although suppressive ART is allowing PLWH to achieve normal or near normal life spans, this is not necessarily accompanied by a normal health span or a healthy aging . Indeed, HIV persistence is associated with a chronic immune activation and inflammation linked to an increased secretion of pro-inflammatory cytokines. On the other hand, a persistent state of inflammation exacerbates damage in tissues, such as the gastrointestinal tract, resulting in microbial translocation, which further increases inflammation. This persistently activated immunological status predisposes PLWH to develop non-AIDS defining diseases, which correspond to affections related to immunosenescence and therefore, mostly observed in the aging population. Indeed, persistent HIV infection and long-term ART treatment have been associated with the development of metabolic syndrome, cardiovascular diseases, type 2 diabetes, neurocognitive disorders, amongst others. As such, inflammatory markers associated with monocyte and macrophage activation such as IL-6, sCD14, and sCD163 are highly predictive for the development of non-AIDS defining diseases further stressing the important roles of these cells in HIV infection and pathogenesis. In addition, HIV infection and persistence in the central nervous system, particularly in microglia, is associated with the development of HIV-associated neurocognitive disorders (HAND), which occurs in approximately 50% of the HIV+ patients despite suppressive ART. Although the molecular and cellular basis are far to be fully understood, there is evidence showing that persistent immune activation and chronic inflammation in PLWH results from the combination of different conditions including dysbiosis and microbial translocation, co-infections, HIV replication and production. It has been reported that early during infection, HIV attacks the mucosal gut generating a strong depletion of memory CD4+ T-cells and the disruption of the intestinal epithelium, triggering both dysbiosis and the release of bacterial components to the circulation through microbial translocation. As such, the evidence suggests that PLWH possesses an altered intestinal microbiota with increased pro-inflammatory (e.g., Prevotella) and decreased anti-inflammatory bacteria (e.g., Bacteroides) when compared to healthy controls. Moreover, the LPS from translocated Gram-negative bacteria binds to CD14 both soluble or present in the surface of monocytes and macrophages, triggering a strong immune activation through TLR4 and the production of pro-inflammatory cytokines such as IL-6, IL-1β, TNF-α, amongst others. A persistent state of immune activation and inflammation in PLWH is also supported by co-infections with other viruses, including hepatitis C and B viruses (HCV and HBV), cytomegalovirus (CMV), Epstein-Barr virus (EBV) and human papilloma virus (HPV). For instance, some studies have reported that HIV/HCV co-infected patients present higher levels of pro-inflammatory markers including IL-6 and sCD14 when compared with mono infected individuals. Moreover, CMV infection has widely been shown to contribute to HIV infection and persistence at least by promoting bacterial translocation and inflammation in the gut, which attracts HIV target cells, and by promoting inhibitory immune pathways, such as cellular exhaustion or PD-L1 and IL-10 secretion, which favor the survival of HIV-infected cells. Tissue-resident macrophages, including alveolar macrophages in the lung, microglia in the central nervous system or urethral macrophages in the urethra, can serve as long-term reservoirs for the virus, being proposed as key players of HIV-associated pathogenesis. Indeed, macrophages harboring HIV DNA, RNA, proteins, and intact viruses have been detected in patients under suppressive ART. Interestingly, the presence of cell-associated HIV RNA but not the size of intact proviruses has been associated with systemic inflammation, suggesting that viral transcription and HIV RNA metabolism(which are not targeted by ART) are important drivers of immune activation and inflammation. Since none of the current ART drugs target viral RNA metabolism (transcription, processing, or nuclear export), the continuous expression and cytoplasmic accumulation of the HIV RNA in cells from the reservoir might be a major contributor to myeloid cells activation perpetuating chronic inflammation in PLWH despite suppressive ART. Hyperactivation of B-cells induced by pro-inflammatory cytokines is characterized by hypergammaglobulinemia, increased polyclonal B-cell activation, increased cell turnover, expression of activation markers (CD70, CD71, CD80 and CD86), increased differentiation to plasmablast cells, increased production of autoantibodies and an increase in the frequency of B-cell malignancies. The current advances in next generation sequencing technologies has enabled the assessment of the full set of V(D)J rearrangement of the immunoglobulin genes, also known as the B-cell repertoire. A recent study detected shifts in the V gene family usage, higher degrees of somatic hypermutations, and longer heavy chains (CDRH3s) in antibodies of PLWH. However, the role of repertoire divergences and whether it is influenced by the presence of other non-AIDS defining diseases such as metabolic syndrome remains largely unexplored .Metabolic syndrome is defined as having at least three of five components: elevated waist circumference (≥ 88 cm for women, 102 cm for men), elevated triglycerides (≥ 150 mg/dL) or drug treatment for elevated triglycerides, low HDL cholesterol (≤ 40 mg/dL for men, 50 for women) or drug treatment for low HDL; elevated blood pressure (systolic ≥ 130 mm Hg or diastolic ≥ 85 mm Hg) or hypertensive drug treatment, and elevated fasting glucose (≥100 mg/dlL) or drug treatment for elevated glucose. Metabolic syndrome is associated with a poor clinical outcome as it doubles the risk for developing cardiovascular diseases (CVD) and quintuples the risk for the development of type 2 diabetes in the 5 to 10 years after CVD diagnosis. Adults, from the general population, with components of metabolic syndrome are twice as likely to die of a cardiovascular event as those without the syndrome, regardless of a previous history of CVD. Prevalence of metabolic syndrome in PLWH ranges from11 to 48% although it is still uncertain whether this prevalence is higher in PLWH than in the general population. Since adipocytes constitutively secrete IL-6 and TNF-a, accumulation of visceral adipose tissue is one of the major body components contributing to systemic inflammation and therefore, it might be an important contributor to chronic inflammation in PLWH. Moreover, replication-competent HIV has been isolated from adipose tissue derived CD4+T-cells and adipose tissue stromal vascular cells indicating that adipose tissue corresponds to an important reservoir for the virus. Although T-cells and macrophages within adipose tissue are susceptible to HIV infection, it is still unknown how immune cells are activated in metabolic syndrome associated with HIV infection. According to the last National Health Survey, 40% of the Chilean population has metabolic syndrome and based on our estimations, at least a half of the PLWH visiting our centers is suffering from the same health condition. Unfortunately, there is no evidence from Chile regarding critical aspects conditioning the quality of life of PLWH including the immune and inflammatory status, the viral reservoir and how they, together with metabolic syndrome, dictate the clinical outcome of the patients.Importantly, the unhealthy aging associated to the persistent inflammation due to chronic HIV infection is expected to overwhelm health care systems being particularly important in resource-limited countries such as Chile.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria will be considered in the adult cohort:

* Adults over 18 years
* Signed informed consent
* HIV diagnosis confirmed by the Public Health Institute
* Patients under clinical control in any of the participating centers
* Availability to attend the taking of samples and medical controls

The following inclusion criteria will be considered in the pediatric cohort:

* Infants and children younger 18 years
* Patients under control in any of the participating center
* Signed informed consent by parents or legal guardians of the minor. In children 8 years and older, also informed assent
* In infants under 4 months of life, HIV diagnosis by a first positive RT-PCR for HIV performed at the Public Health Institute. In infants and children over 4 months, HIV diagnosis is confirmed by the Public Health Institute.
* Children exposed to HIV during pregnancy, labor or breastfeeding of mothers with confirmed HIV, with a negative diagnosis.
* Availability to attend the taking of samples and medical controls, and without medical contraindications for taking the samples (severe anemia according to age).

The following exclusion criteria will be considered in both cohorts:

- The only exclusion criterion will be the patient's refusal to participate in the case of adults and in the case of minors, the non-signature of the informed consent by the legal guardians and the minor's non-assent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be obtained from different centers from Santiago and Punta Arenas, including Fundación Arriarán, Hospital Clínico de Magallanes, Hospital del Salvador. These cohorts include men and women, from adolescence to adulthood and senior patients living with HIV under suppressive ART and presenting or not metabolic syndrome.
  A group of HIV negative individuals with and without metabolic syndrome will also be invited to participate to be used as controls when required.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Characterization of a Chilean cohort of PLWH with and without metabolic syndrome. | 12 month

SECONDARY OUTCOMES:
Sociodemographic data questionnaire | 12 months
  Number of illnesses, medical treatments, vaccination records, metabolic syndrome status, quality of life, and informed consent.
Dysbiosis by NGS | 12 months
  Taxonomic frequency.
Dysbiosis by NGS | 12 months
  Diversity index.
Immune cell repertoire by Flow Citometry | 12 months
  Absolute count of T cells.
Immune cell repertoire by Flow Citometry | 12 months
  Relative count of T cells.
Immune cell repertoire by Flow Citometry | 12 months
  Relative count of Memory T cells
Immune cell repertoire by Flow Citometry | 12 months
  Relative count of Naive T cells.
Immune cell repertoire by Flow Citometry | 12 months
  Relative count of Follicular helper T cells.
Immune cell repertoire by Flow Citometry | 12 months
  Relative count of Regulatory T cells (Tregs).
Immune cell repertoire by Flow Citometry | 12 months
  Relative count of Th17 cells.
Immune cell repertoire by Flow Citometry | 12 months
  Relative count of CD8⁺ activated T cells.
B-cell receptor repertoire by NGS | 12 months
  VDJ family rearrangement frequency
Immune cell repertoire by NGS | 12 months
  Clonal abundance.
Immune cell repertoire by NGS | 12 months
  Diversity index (Shannon, Hill, Gini).
B-cell receptor repertoire by NGS | 12 months
  CDR3 characterization (size, physicochemical composition).
Single-cell RNA by scRNA-seq | 18 months
  Expression levels
Single-cell RNA by scRNA-seq | 18 months
  Clonotype characterization
Proteomics by Mass spectrometry | 18 months
  Identification and quantification of proteins
Proteomics by Mass spectrometry | 18 months
  Differential expression of proteins Mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Soto-Riffo, PhD, Principal Investigator — University of Chile
Locations (1):
- Centro Asistencial Docente y de Investigación, Universidad de Magallanes, Punta Arenas, Punta Arenas, Chile

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared is all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following the data is cleaned, quality checked, and analyzed, the data will be available to the general research community. All data made available for public use will be de-identified data, i.e., stripped of private, protected health information that could be used to deduce the identity of individual subjects, in compliance with the rule.
Access Criteria: InflammAIDS website will display the data and statistical analysis.
URL: https://chair.med.uchile.cl

REFERENCES:
- [Background] Giraldo-Ocampo S, Valiente-Echeverria F, Soto-Rifo R. Host RNA-Binding Proteins as Regulators of HIV-1 Replication. Viruses. 2024 Dec 31;17(1):43. doi: 10.3390/v17010043. PMID 39861832
- [Background] Acevedo ML, Gaete-Argel A, Alonso-Palomares L, de Oca MM, Bustamante A, Gaggero A, Paredes F, Cortes CP, Pantano S, Martinez-Valdebenito C, Angulo J, Le Corre N, Ferres M, Navarrete MA, Valiente-Echeverria F, Soto-Rifo R. Differential neutralizing antibody responses elicited by CoronaVac and BNT162b2 against SARS-CoV-2 Lambda in Chile. Nat Microbiol. 2022 Apr;7(4):524-529. doi: 10.1038/s41564-022-01092-1. Epub 2022 Apr 1. PMID 35365787
- [Background] Gonzalez-Puelma J, Aldridge J, Montes de Oca M, Pinto M, Uribe-Paredes R, Fernandez-Goycoolea J, Alvarez-Saravia D, Alvarez H, Encina G, Weitzel T, Munoz R, Olivera-Nappa A, Pantano S, Navarrete MA. Mutation in a SARS-CoV-2 Haplotype from Sub-Antarctic Chile Reveals New Insights into the Spike's Dynamics. Viruses. 2021 May 11;13(5):883. doi: 10.3390/v13050883. PMID 34064904